CLINICAL TRIAL: NCT06228950
Title: Effectiveness of Mindfulness-Based Intervention for Emotional and Behavioural Problems of Students With Visual Impairment
Brief Title: Mindfulness-Based Intervention for Emotional and Behavioural Problems of Students With Visual Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Tehmeena Hanif, Principal Investigator, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FJWU/EC/2023/65
Record Dates: First submitted 2024-01-07; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Emotional Problem; Behavior Problem
Keywords: Emotional and Behavioural Problems Mindfulness Students
MeSH Terms: conditions — Mental Disorders | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT) design will be used in this interventional study to evaluate the effectiveness of mindfulness-based intervention for emotional and behavioral problems of students with visual impairment. Participants in RCT will be randomized in the intervention and the control group. Urdu-translated and adaptive mindfulness-based intervention that is MBSR designed specifically to meet the needs of students with visual impairment will be given to the intervention group. The MBSR training program consisted of 8-week group sessions with a duration of 50 to 90 minutes each for a group of 5-8 members. The intervention will include a body scan, sitting meditation, yoga, breathing exercises, guided mindfulness exercises, loving kindness etc to improve emotional and behavioral problems. Standardized measures will be used to evaluate changes in pre and post-intervention.
Who Masked: Participant, Investigator
Masking Description: Double-Blind, neither the participant nor the investigator know what they are getting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A structured MBSR training for this study will be given to the intervention group of students with visual impairment. The intervention will include body scan, sitting meditation, yoga, breathing exercises, guided mindfulness, loving kindness, etc exercises to improve the emotional and behavioural problems of students with visual impairment.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Wait-list Control Group (No Intervention): The Wait-list control group will receive no intervention. This group will serve as a comparison group to evaluate the specific effect of the mindfulness based intervention.

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — A therapeutic approach called mindfulness-based stress reduction, or MBSR, aims to reduce emotional and behavioral problems by fostering mindfulness, which is an impartial awareness of the present moment. MBSR will be an 8-week training course for students with visual impairment. MBSR training, translated and adapted in Urdu language that includes 8 audios and worksheets corresponding to each week. Worksheets to record home practice will be filled upon receiving oral feedback from the students with visual impairment. Face-to-face group-based sessions will be conducted weekly.
  Arms: Intervention Group

SUMMARY:
Current study will be conducted on the Effectiveness of Mindfulness-Based Intervention for Emotional and Behavioural Problems of Students with Visual Impairment. Mindfulness-based Intervention that is Mindfulness-Based Stress Reduction (MBSR) will be used in the current study which is adapted and translated in Urdu language; the pilot trial of MBSR will be conducted after adaptation and translation.

The present study will be conducted in two phases

* First phase of the study would be a cross-sectional survey in which the researcher will conduct a baseline assessment to identify psychosocial predictors such as psychological distress, parental acceptance and rejection, social support, and mindfulness which are associated with the emotional and behavioural problems of students with visual impairment. Further emotional and behavioural problems of the students with visual impairment will identify.
* The second phase of the research would be a Randomized Controlled Trial in which students with Visual Impairment who has scored high on psychosocial predictors and emotional & behavioural problems would be randomly assigned to intervention & control groups to get the MBSR training. After the successful training post-assessment would be conducted to check the efficacy of MBSR.
* The current study will be conducted in Rawalpindi Islamabad after obtaining permission from the relevant authorities.
* Data would be collected from the students with visual impairment and their respective parents.

DETAILED DESCRIPTION:
The study is designed to assess the Emotional and Behavioural Problems (EBPs) of Students with Visual Impairment studying at special education schools for impaired vision and to evaluate the relationship between the scores of psychosocial predictors that are associated with EBPs and selected demographic variables of these students. According to a literature review among all types of disabilities, a high occurrence of psychological disorder was found in VI children. So, the present study aimed to assist students with visual impairment in controlling the occurrence of different emotional and behavioural problems. Additionally, the current study will be advantageous for instructors, coaches, and policymakers to consider the role of educational psychologists in special school settings. Visual impairment can cause problems in daily life, but a person with sound mental health can better deal with it. So, the present study will contribute a lot to society by improving the life quality of these special children. Students with visual impairment in their school settings will utilize the practice of MBSR to reduce stress and to increase their emotional and adaptive behaviours. The purpose of current research is to integrate mindfulness practices in special school settings to provide the behavioural support for adolescents with visual disabilities so that they can be more successful both socially and academically.

Sample The present study will be conducted with students who will be Visually Impaired (partial or complete). Data will also be collected from their respective parents. The sample will be taken from different schools of blinds, centers, and special schools in Rawalpindi/Islamabad. The age group of samples will range from 13 to 17 years. Purposive sampling will be used and those participants will be selected who will be available and volunteer to participate at the time of data collection. Data will be collected in one-on-one interviews by oral administration of questionnaires.

MBSR will be translated and adapted into Urdu language. Permission to translate into Urdu language will be taken from the relevant authority. In the first phase, participants will be initially asked about demographic variables. The researcher would identify the psychosocial predictors of emotional and behavioural problems of students with Visual Impairment based on the scores of Depression Anxiety Stress Scale-21 (DASS-21), Parental Acceptance and Rejection Questionnaire (Child PARQ), Multidimensional Scale of Perceived Social Support (MSPSS) and Mindfulness Attention Awareness Scale-Adolescents (MAAS-A). Further emotional and behavioural problems of the students with visual impairment will identify by SDQ Self and SDQ Parent report form scores. Participants will be assured about the confidentiality of the data and its findings that will only be used for the cause of the research project.

In the second phase cohort would be identified from the participants who would score high on DASS-21, Child PARQ, SDQ Self, and SDQ Parent report form and low on MSPSS & MAAS-A. They would be screened out as potential cohorts for Randomized Control trials (RCT). Participants would be randomly assigned to interventional and control groups by using the random number method. Participants who would be assigned to the interventional group will be exposed to the Urdu-translated and adapted Mindfulness-Based Stress Reduction (MBSR) training. Students who would be assigned to the interventional group will receive 8 weeks of therapeutic intervention however the students who are randomly assigned to the control group will be given no intervention. The MBSR training program consisted of 8-week group sessions with a duration of 50 to 90 minutes each. Each week will focus on a particular theme related to the emotional and behavioural problems of students with Visual Impairment. After the successful completion of 8 weeks of MBSR training both groups will appear for post-assessment. The same aforementioned measures will be used in post-assessment.

ELIGIBILITY:
Inclusion Criteria:

* Parents and their children who will be in the age range of at least 13-17 years will be included in the present study. All students who will participate in this study will be partially or completely visually impaired.
* Participants who scored higher on DASS-21, PARQ, SDQ self, and SDQ parent report form and low on MSPSS and MAAS-A in phase I will be included in phase II of the study i.e. Randomized Control Trial.

Exclusion Criteria:

* Exclusion criterion will be; students and parents who would not be willing to participate and who refuse to give consent. Other disabilities in students will not be considered (e.g. hearing disability or other physical disabilities).
* Participants who have gone through critical medical conditions like psychological treatment or surgery or have co-morbid problems would be excluded.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Strength and Difficulties Questionnaire (Self Report Version) | 2 Months
  It has 25 items, with subscales that generate scores for emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behaviour. It is a 3-point Likert-type scale. The Self Report Version score ranges from minimum to maximum which is 0 to 50. Low scores indicate better outcomes and high scores indicate worse outcomes which is high Emotional and Behavioural Problems in students with visual impairment.
Strength and Difficulties Questionnaire (Parent Report Version) | 2 Months
  It has 25 items that measures the same attributes as the self-report version. It is a 3-point Likert type scale. The Parent Report Version score ranges from minimum to maximum which is 0 to 50. Low scores indicate better outcomes whereas high scores indicate worse outcomes that is high Emotional and Behavioural Problems in students with visual impairment.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale-21 | 2 Months
  Depression Anxiety Stress Scale-21 is a comprehensive measure for depression, anxiety, and stress. it is a four-point Likert-type scale. The score ranges from minimum to maximum which is 0 to 63. Low scores indicate better outcomes whereas high scores indicate worse outcomes that is high Psychological Distress.
Child Parent Acceptance-Rejection Questionnaire | 2 Months
  It is a self-report measure to identify perception of individual about the parental treatment that he/she received during childhood. It has four subscales that are Warmth/Affection, Hostility/Aggression, Indifference/Neglect, and Undifferentiated rejection. It has two versions; mother and father. Each consists of 24 items on a 4 point Likert-type scale. The score range of the scale from minimum to maximum is 24 to 96. Low scores indicate the better outcome which is the lowest rejection and highest acceptance whereas high scores indicate the worse outcome which is the highest rejection and lowest acceptance.
Multidimensional Scale of Perceived Social Support | 2 Months
  It is a self-report inventory which is used to assess persons' perception of social support that they receive from the family, friends or significant others in stressful situations. It contains 12 items with 7 point likert type scale. The score range of the scale from minimum to maximum is 12 to 84. Low scores indicate a worse outcome that is low level of perceived social support whereas as high score indicate better outcome.
Mindfulness Attention Awareness Scale-Adolescents | 2 Months
  It is a 14-item scale measuring the development of mindfulness. The score range of the scale from minimum to maximum is 14 to 84. Low scores indicate a worse outcome that is low level of mindfulness whereas a high score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tehmeena Hanif, PhD Scholar, Principal Investigator — Fatima Jinnah Women University Rawalpindi Pakistan
Locations (1):
- Tehmeena Hanif, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No